CLINICAL TRIAL: NCT02983123
Title: Introduction of an 1-hour Algorithm for High-sensitivity Cardiac-specific Troponin T for Faster Assessment of NSTEMI in a Low-prevalence Population at Oslo Accident and Emergency Outpatient Clinic
Brief Title: One-hour Troponin in a Low-prevalence Population of Acute Coronary Syndrome
Acronym: OUT-ACS
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Principal Investigator, Dan Atar, Professor of Cardiology and Head of Research, Oslo University Hospital
Other Study IDs: 2016/1241/REK; 2016/13308 (Other: PVO OUS)
Record Dates: First submitted 2016-11-29; First posted 2016-12-06 (Estimated); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Non-ST Elevation Myocardial Infarction; Acute Coronary Syndrome; Angina, Unstable; NSTEMI - Non-ST Segment Elevation MI
Keywords: Acute MI; Acute myocardial infarction cardiac troponin; High-sensitivity cardiac troponin T; 0/1-hour algorithm; Outpatient clinic; Cardiac troponin; Chest pain
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction; Acute Coronary Syndrome; Angina, Unstable; Chest Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1 hour-troponin: 1-hour troponin collected of all recruited patients in addition to the daily routine with serial troponins collected at 0- and 4/6 hours.
  Interventions: Procedure: 1-hour hs-cTnT

INTERVENTIONS:
Procedure: 1-hour hs-cTnT

SUMMARY:
This study aims to evaluate if the 1-hour rule-in/rule-out algorithm for a high-sensitivity cardiac troponin T (hs-cTnT) is safe and effective for use in the primary care where the patients have a lower pretest probability of an acute myocardial infarction (MI). During this study troponins will be collected at 0-, 1- and 4/6-hours, where absolute changes in the values will decide whether the patient need hospitalization or not.

DETAILED DESCRIPTION:
Many patients seek Oslo Accident and Emergency Outpatient Clinic (OAEOC) with chest pain. The majority of these patients have symptoms suggestive of a benign non-cardiac chest pain. These patients do not need a directly transfer to the hospital, but can be admitted to the Observation Unit at the OAEOC for further pre-hospital testing, including serial troponins for a safe rule-out of acute MI. The main goal of this study is to improve the current routine at the Observation Unit at OAEOC by introducing the 1-hour algorithm for hs-cTnT for a faster rule-in/rule-out of acute MI.

All recruited patients will have serial troponins drawn at 0, 1- and 4/6 hours, with the main hypothesis that the absolute changes within 1 hour can be used as surrogates for the changes and conclusions drawn after 4/6 hours. The cut-off levels used within the 0/1-hour algorithm are assay specific as specified in the 2015 European Society of Cardiology Guidelines for the management of acute NSTEMI.

ELIGIBILITY:
Inclusion Criteria:

* Patients at the outpatient clinic with suspected non-cardiac chest pain/symptoms who need further testing for a safe rule-out of an acute MI
* Written informed consent

Exclusion Criteria:

* Acute STEMI (ST-elevation myocardial infarction) (directly to the hospital)
* Strong suspicion of an acute NSTEMI/unstable angina (directly to the hospital)
* Terminal kidney disease with a glomerular filtration rate (GFR) < 30
* Unable to communicate in Norwegian, Swedish, Danish or English language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the Oslo Accident and Emergency Outpatient Clinic with symptoms suggestive of a benign non-cardiac chest pain, who needs further pre-hospital testing at the Observation Unit for a safe rule-out of an acute MI.
Sampling Method: Non-Probability Sample
Enrollment: 1750 (Actual)
Dates: Start 2016-11-15 (Actual); Primary Completion 2018-10-22 (Actual); Study Completion 2018-10-22 (Actual)

PRIMARY OUTCOMES:
Number of patients transferred to the hospital (rule-in) according to the 1-hour algorithm | 7-10 hours
  The troponin tests will be sent to the laboratory for analysis every 4th hour. The tests are analyzed in 1-2 hours.
Number of patients without significant changes (rule-out) according to the 1-hour algorithm | 7-10 hours
  The troponin tests will be sent to the laboratory for analysis every 4th hour. The tests are analyzed in 1-2 hours.

SECONDARY OUTCOMES:
Number of patients with significant change in the 3rd troponin (drawn after 4-6 hours) who were not identified by the 1-hour algorithm | 10 hours
Significant changes between the first and second ECG? | 6 hours
Number of patients with NSTEMI admitted to the hospital from the Observation Unit at the OAEOC | 1 week
  The final diagnosis will be collected from all patients who were admitted to the hospital from the Observation Unit during the study
90 days follow-up of all recruited patients | 90 days
  How many will have an acute MI the next 3 months?

CONTACTS AND LOCATIONS:
Overall Officials: Dan Atar, MD, PhD, Study Director — Oslo University Hospital and University of Oslo, Norway
Locations (1):
- Oslo Accident and Emergency Outpatient Clinic, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Johannessen TR, Melessen IMB, Vallersnes OM, Manten A, Halvorsen S, Atar D, Harskamp RE. Adequately identifying low-risk chest pain in emergency primary care: evaluating the performance of preHEAR(T) based on two European cohorts. Open Heart. 2025 Jul 27;12(2):e003362. doi: 10.1136/openhrt-2025-003362. PMID 40716792
- [Derived] Johannessen TR, Halvorsen S, Atar D, Vallersnes OM. Performance of the Novel Observation Group Criteria of the European Society of Cardiology (ESC) 0/1-Hour Algorithm in a Low-Risk Population. J Am Heart Assoc. 2022 Apr 5;11(7):e024927. doi: 10.1161/JAHA.121.024927. Epub 2022 Mar 30. No abstract available. PMID 35352564
- [Derived] Johannessen TR, Atar D, Vallersnes OM, Larstorp ACK, Mdala I, Halvorsen S. Comparison of a single high-sensitivity cardiac troponin T measurement with the HEART score for rapid rule-out of acute myocardial infarction in a primary care emergency setting: a cohort study. BMJ Open. 2021 Feb 24;11(2):e046024. doi: 10.1136/bmjopen-2020-046024. PMID 33627355
- [Derived] Johannessen TR, Vallersnes OM, Halvorsen S, Larstorp ACK, Mdala I, Atar D. Pre-hospital One-Hour Troponin in a Low-Prevalence Population of Acute Coronary Syndrome: OUT-ACS study. Open Heart. 2020 Jul;7(2):e001296. doi: 10.1136/openhrt-2020-001296. PMID 32719074